CLINICAL TRIAL: NCT00397878
Title: Phase II Study of AZD0530 (NSC 735464) in Patients With Previously Treated Metastatic Colorectal Cancer
Brief Title: AZD0530 (NSC 735464) in Treating Patients With Previously Treated Metastatic Colon Cancer or Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after all enrolled participants progressed.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00067; NCI-2013-00067 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000512970; MDA-2005-0977; NCI-7569; 2005-0977 (Other: M D Anderson Cancer Center); 7565 (Other: CTEP); N01CM62202 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-07

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — saracatinib

ARMS (1):
- Treatment (saracatinib) (Experimental): Patients receive oral AZD0530 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: saracatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: saracatinib — Given orally
  Other Names: AZD0530
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well AZD0530 works in treating patients with previously treated metastatic colon cancer or rectal cancer. AZD0530 may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival (PFS) at 4 months in metastatic colorectal carcinoma patients receiving daily doses of AZD0530.

SECONDARY OBJECTIVES:

I. Evaluate the objective response rate (RR) and overall survival (OS) of patients with metastatic colorectal cancer who are treated with AZD0530.

II. In patients who consent, both blood and tissue samples will be collected for laboratory correlates. Assess in a preliminary manner the association between correlative markers and the potential downstream effects of AZD0530 on IL-8, VEGF, specific Src-regulated markers in focal adhesions, adherens junctions, and angiogenesis on clinical outcome in pre- and post-treatment tumor samples.

OUTLINE:

Patients receive oral AZD0530 once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic
* Patients must have measurable disease, defined (per RECIST criteria) as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or >= 10 mm with spiral CT scan
* Patients must have received one and only one prior chemotherapy regimen for metastatic colorectal cancer; patients may have received biologic therapy (e.g., bevacizumab) in combination with chemotherapy as part of their prior chemotherapy
* ECOG performance status 0-2
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional ULN
* AST(SGOT)/ALT(SGPT) =< 3.0 x institutional ULN
* Creatinine within normal institutional limits OR estimated CrCl (Cockcroft-Gault) or 24 hr urine collection of >= 50 mL/min
* The effects of AZD0530 on the developing human fetus at the recommended therapeutic dose are unknown; however, AZD0530 has been shown to cause gross fetal malformations and to negatively impact embryo fetal survival in rats; for this reason and because many tyrosine kinase inhibitors are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and up to 30 days following removal from the study; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; women of child-bearing potential will have serum beta-Hcg levels drawn up to 7 days prior to receiving study treatment
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD0530, breastfeeding should be discontinued if the mother is treated with AZD0530
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to study registration or those who have not recovered from treatment related adverse events > grade 1 (except for neuropathy [ies] which may be =< grade 2) due to agents administered more than 4 weeks earlier
* Use of specifically prohibited CYP3A4-active agents or substances are not permitted during protocol treatment, and patients who must continue treatment with these agents are not eligible; prohibited drugs should be discontinued seven (7) days or 5 half-lives (whichever is the longer time period) prior to the administration of the first dose of AZD0530 and for 7 days or 5 half-lives (which ever is the longer time period) following discontinuation of AZD0530
* Patients may not be receiving any other investigational agents
* Patients with greater than +1 proteinuria on two consecutive readings taken no less than 24 hours apart are ineligible
* Patients with QTc prolongation (defined as a QTc interval greater than or equal to 480 msecs) are ineligible
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (requiring parenteral antibiotics at the time of registration), cardiac disease NYHA class III or IV, unstable angina pectoris, unstable cardiac arrhythmia or tachycardia (heart rate >= 100 beats per minute), poorly controlled hypertension (systolic blood pressure >= 140 mmHg or diastolic blood pressure >= 90 mmHg)
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow AZD0530 tablets are excluded
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Pregnant women are excluded from this study because AZD0530 has the potential for teratogenic or abortifacient effects as shown by the gross fetal malformation and effects on embryofetal survival seen in reproductive toxicity studies in the rat
* Patients with a history of another primary malignancy within the last 5 years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix
* Patient who are known to be HIV-positive are ineligible because of the potential for pharmacokinetic interactions with AZD0530 and antiretroviral therapy (HAART)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Eng, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: November 16, 2006 to April 08, 2008. Recruitment done at University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Treatment (Saracatinib): Oral AZD0530 175 mg once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Saracatinib)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Time period of metastatic colorectal patients with one previous chemotherapy treatment for metastatic disease who are alive and progression free after commencing the experimental therapy. A 95% posterior credible intervals used.
Time Frame: Time from start of treatment to time of progression, up to 4 months
Measure: Median (Full Range); unit: weeks
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 10
weeks | 7.9 [2.1 to 9.6]

2. Secondary Outcome: Overall Survival
Description: Number of participants who survived up to 5 years
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 10
Participants | 6

3. Secondary Outcome: Time to Progression
Description: Number of participants who progressed on treatment within less than or equal to 2 cycles (cycle=28 days; within 54 days PD).
Time Frame: within 54 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 10
Participants | 10

4. Other Pre Specified Outcome: Pre- and Post-treatment Expression Values for Each Biological Correlate
Description: Statistical significance of the associations assessed using a nonparametric Sign Test performed on the difference of the post-treatment and pre-treatment values. A two-sided .05 significance level to be used.
Time Frame: Up to 2 weeks
Population: No patients consented to optional tissue analysis.
Arm/Group | Treatment (Saracatinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected while participant was receiving treatment and up to 30 days after the last dose of treatment. Total study period was from January 10, 2007 to February 25, 2009.
Arm/Group | Treatment (Saracatinib)
Serious Adverse Events (participants affected / at risk) | 9/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=10)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 1 (1)
Death NOS (General disorders) | 6 (10)
Dehydration (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (6)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Saracatinib) (N=10)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 8 (12)
Anorexia (Gastrointestinal disorders) | 5 (5)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) — Ascites
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 9 (12)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood bilirubin increased (Hepatobiliary disorders) | 3 (3)
Cholesterol high (Metabolism and nutrition disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (8)
Creatine phosphokinase (CPK) increased (Metabolism and nutrition disorders) | 1 (1)
Creatinine increased (Metabolism and nutrition disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Extraocular muscle paresis (Musculoskeletal and connective tissue disorders) | 1 (1)
Fatigue (General disorders) | 10 (16)
Fever (General disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4)
Hypertension (Cardiac disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (11)
Hypothyroidism (Endocrine disorders) | 1 (1)
Immune system disorders (Immune system disorders) | 2 (2) — Seasonal allergies
Urinatry Tract Infections (Infections and infestations) | 5 (6)
Insomnia (Psychiatric disorders) | 2 (2)
Elevated Blood Counts (Investigations) (Infections and infestations) | 5 (6) — LOW CHLORIDE, ELEVATED Blood urea nitrogen (BUN), ELEVATED URIC ACID, ELEVATED lactate dehydrogenase (LDH) and URINE KETONES
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (8)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Platelet count decreased (Blood and lymphatic system disorders) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Repiratory, Running Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Tumor pain (General disorders) | 2 (2)
Urinary frequency/retention (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (6)
Watering eyes (Eye disorders) | 2 (2)
Weight loss (General disorders) | 2 (2)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less